CLINICAL TRIAL: NCT05160493
Title: The Effect of Esketamine Combined With Pregabalin on Chronic Postsurgical Pain in Patients After Craniotomy.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20211206
Record Dates: First submitted 2021-12-07; First posted 2021-12-16 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Chronic Postsurgical Pain
Keywords: Esketamine; Pregabalin; Craniotomy; Chronic Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Esketamine; Pregabalin; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-ketamine and pregabalin (Experimental): Drug: S-ketamine and pregabalin
  * Drug: Pregabalin 150mg (2hrs) pre operatively and 75mg twice daily post operatively for 7 days(POD1-7),followed by dose reduction to 75mg once daily for 7days(POD8-14)
  * Drug: S-ketamine infusion 0.5 mg/kg bolus after induction of anesthesia +0.12 mg/kg/h continuous intravenous infusion for 48 h
  Interventions: Drug: S-ketamine and pregabalin
- Normal saline and placebo capsule (Placebo Comparator): Drug: Normal saline and placebo capsule
  * Drug: Placebo capsules :Two placebo capsules(2hrs) preoperatively and twice daily post operatively for 7days, followed by dose reduction to single capsule once daily for 7days
  * Drug: Normal saline• 0.9% saline bolus after induction of anesthesia +intravenous infusion for 48 hours
  Interventions: Drug: Normal saline and placebo capsule

INTERVENTIONS:
Drug: S-ketamine and pregabalin — S-ketamine and pregabalin
  * Drug: Pregabalin • 150mg (2hrs) pre operatively and 75mg twice daily post operatively for 7 days(POD1-7),followed by dose reduction to 75mg once daily for 7days(POD8-14)
  * Drug: S-ketamine infusion • 0.5 mg/kg bolus after induction of anesthesia +0.12 mg/kg/h continuous intravenous infusion for 48 h
  Arms: S-ketamine and pregabalin
Drug: Normal saline and placebo capsule — Normal saline and placebo capsule
  Arms: Normal saline and placebo capsule

SUMMARY:
Chronic postsurgical pain (CPSP), which is one of the most common and serious long term complication of surgery，occurs in approximately 10% of patients after a surgical procedure. Craniotomy was previously considered to have less chronic pain than other surgical procedures. Contrarily, studies have reported incidences of chronic headache varies for type of craniotomy, ranging from 23% to 34% at three months and 12% to 16% at one year after surgery. In addition，CPSP is associated with adverse events, including postoperative morbidity, increased health-care costs, significant impaired on quality of life, prolonged opioid use. Optimising perioperative pain management should reduce the incidence of CPSP; The non-opioid analgesics, such as ketamine and pregabalin, have also been used as components of multimodal anesthetic protocols. Postoperative pain scores and opioid use are significantly reduced in thoracotomy surgical patients given ketamine and pregabalin compared to control groups.however, there is currently a lack of evidence regarding which therapeutic options are most effective in reducing the incidence of chronic post-craniotomy headache. The investigators hypothesis is that sketamine combined with pregabalin reduces significantly chronic postoperative pain after craniotomy and improves patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age ≥18 years, male or female
* American Society of Anaesthesiology (ASA) status I-III
* Patients undergoing elective craniotomy

Exclusion Criteria:

* Patients unable to complete scale assessment
* Pregnant or lactating women
* Patients with preoperative chronic pain syndrome
* Patients with previous craniotomy history
* Patients with a history of mental illness who are receiving medication
* Patients with liver and kidney dysfunction
* Patients have taken pain medication within two weeks
* Patients with history of adverse reactions to pregabalin, ketamine and esticketamine
* Patients with history of drug abuse;
* BMI>35.0 kg · m - 2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Proportion of craniotomy patients with NRS score greater than one 3 months after surgery | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph D., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided